CLINICAL TRIAL: NCT01123850
Title: A Prospective Study Assessing Clinical Outcomes and Radiographic Results After the Use of CopiOs(R) Bone Void Filler (BVF)Sponge in a Posterolateral Fusion Procedure (PLF).
Brief Title: CopiOs Posterolateral Fusion Procedure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-001
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Spondylolisthesis; Stenosis
Keywords: CopiOs; Degenerative spondylolisthesis,; stenosis with instability, or; degenerative disc disease as diagnosed by radicular signs and/or imaging studies
MeSH Terms: conditions — Spondylolisthesis; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single ARM - Copios Bone Filler (Active Comparator): All subjects will undergo an instrumented, pedicle screw PLF procedure. Autograft or other interbody devices identified by the surgeon to be in the best interest of the patient may be used. Enrolled patients will receive CopiOs BVF sponge soaked with bone marrow aspirate on one side and autologous bone on the other side. All patients will receive both CopiOs BVF and autologous bone. Patients will serve as self-controls in this counter-balanced study.
  Interventions: Device: Copios

INTERVENTIONS:
Device: Copios — Bone Void Filler

SUMMARY:
To compare radiographic data collection from patients undergoing instrumented PLF with CopiOs(R) BVF or instrumented PLF with autologous bone and to assess overall clinical outcomes. Patients will serve as self controls.

DETAILED DESCRIPTION:
This is a prospective, counter-balanced study involving 85 subjects at up to 8 investigative centers. Each subject will be an appropriate candidate for an instrumented PLF and will meet the inclusion and exclusion criteria. All subjects will undergo an instrumented, pedicle screw PLF procedure. Autograft or other interbody devices identified by the surgeon to be in the best interest of the patient may be used. Enrolled patients will receive CopiOs BVF sponge soaked with bone marrow aspirate on one side and autologous bone on the other side. All patients will receive both CopiOs BVF and autologous bone. Patients will serve as self-controls in this counter-balanced study. Data will be collected pre-operatively, operatively and post-operatively at six and twelve months.

The study objectives include: Radiographic success of CopiOs is non-inferior to autograft with clear evidence of bridging bone. Radiographic analysis will be used to show that CopiOs works as well as autograft when comparing the rate of fusion at 6 and 12 months. The CT scan (12 month) will show that CopiOs works as well as autograft when comparing the fusion mass between the transverse processes. Additionally, clinical success will be determined by an improvement of 15 percentage points using the Oswestry Disability Index and maintenance or improvement in the motor and sensory components of the neurological assessment from preoperative to postoperative. Since patients serve as self-controls there will be no clinical success comparisons between the groups. Rather, clinical success will be measured on overall improvement based on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be skeletally mature; between the ages of 21 and 75
* Patients having degenerative spondylolisthesis, stenosis with instability, or degenerative disc disease as diagnosed by radicular signs and/or imaging studies
* Patients will be medically indicated for a single-level, instrumented PLF between L2 and S1 per their surgeon
* Patient must be willing and able to comply with study requirements, including all necessary study related paperwork and follow-up visits

Exclusion Criteria:

* Use of iliac crest bone graft;
* Any previous lumbar spinal surgeries at indicated level;
* Any medical or physical condition that would preclude the potential benefit of spinal surgery;
* Use of a dynamic stabilization systems;
* Sites where stresses on void will exceed the load strength of fixation of hardware;
* Segmental defects;
* Significantly impaired vascularity proximal to the surgical site;
* Sites in direct contact with articular space;
* Soft tissue deficit not allowing closure;
* Active systemic or local infection;
* Severe degenerative bone disease;
* Patients with osteoporosis who are actively under treatment;
* Extreme obesity, as defined by NIH Clinical Guidelines Body Mass Index (BMI>40 kg/m2);
* Active malignancy;
* Patients with a history of multiple allergies;
* Patients with known allergies to bovine collagen;
* Hypercalcemia;
* Pregnancy;
* Mental illness;
* Alcohol or drug abuse;
* Incarceration.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Florida Hospital, Orlando, Florida
  - Neurological Surgery of Southern Illinois, Belleville, Illinois
  - Indiana Orthopedic Center, Indianapolis, Indiana
  - Las Cruces Orthopaedic Associates, Las Cruces, New Mexico
  - Upstate Bone and Joint Center, East Syracuse, New York
  - Scott and White Healthcare, Temple, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single ARM - Copios Bone Filler
Started | 45
Completed | 0
Not Completed | 45
Not completed — Slow enrollment | 45

BASELINE CHARACTERISTICS:
Arm/Group | Single ARM - Copios Bone Filler
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Study was terminated for slow enrollment. Data was not analysed.
  Male | NA — Study was terminated for slow enrollment. Data was not analysed.
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Fusion Assessment
Description: Fusion at 12M using radiograph Fusion Mass at 12M using CT
Time Frame: 6 M, 12 M
Population: Study was terminated due to slow enrollment, there was no data analysis
Arm/Group | Single ARM - Copios Bone Filler
Number analyzed (Participants) | 0

2. Secondary Outcome: Outcome Measure - Pain, Life Quality, Satisfaction
Time Frame: PreOp, Surgery, 6M, 12M
Population: Study was terminated due to slow enrollment, there was no data analysis
Arm/Group | Single ARM - Copios Bone Filler
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Single ARM - Copios Bone Filler
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No